CLINICAL TRIAL: NCT05761522
Title: Cardiac Effects of Norepinephrine After the Initial Phase of Septic Shock
Brief Title: Cardiovascular Effects of Norepinephrine
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PZ23020*
Record Dates: First submitted 2023-02-07; First posted 2023-03-09 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Septic Shock
Keywords: ECHOCARDIOGRAPHY; CARDIAC FUNCTION; NOREPINEPHRINE; SEPTIC SHOCK
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with septic shock for 24 hours or more: Adult patients suffering from septic shock, after 24 hours of their diagnosis. Presenting with Mean arterial pressure (MAP)<65 mmHg or the target MAP For whom the physician in charge decided to increase the norepinephrine dose
  Interventions: Other: transthoracic echocardiography

INTERVENTIONS:
Other: transthoracic echocardiography — * Concerning the main judgment criterion and the secondary judgment criteria:
    * Left ventricular ejection fraction (LVEF) by the Simpson Biplane method,
    * Cardiac output and cardiac index by continuity equation (measurement of left ventricular outflow chamber (mm) and sub-aortic time-velocity integral (cm/s)).
    * Tricuspid Annular Systolic Excursion (TAPSE) (mm)
    * S wave at the tricuspid ring (cm/s)
  * Other parameters collected systematically:
    * Surface of the left ventricle (end-systolic and end-diastolic),
    * Global strain of the left ventricle
    * Mitral Annular Plane Systolic Excursion (MAPSE) (mm)
    * Left ventricular filling pressure (LVRP) (at the mitral annulus, E, A, e', S' waves, E/A ratio, E/e');
    * Maximum tricuspid regurgitation velocity (m/s) to estimate systolic pulmonary arterial pressure (PAPs) (mmHg)

SUMMARY:
Previous studies of our team reported the improvement of myocardial contractility both on hemodynamic parameters (by transpulmonary thermodilution) and morphological (by transthoracic echocardiography: TTE), during the early phase of septic shock (during the first 4 hours management of septic shock).

However, one can wonder about the effect of NAD on myocardial cardiac ouput and contractility beyond the early phase of septic shock, more precisely beyond the first 24 hours. Indeed, while it continues to act on the "stressed" blood volume and the diastolic left ventricular perfusion by increasing the diastolic arterial pressure (DAP), it has been reported in old studies that beyond the early phase, the sensitivity of the β1-adrenergic receptors is altered due to the phenomenon of internalization of these receptors, leading to a reduction of the myocardial response to catecholamines.

The investigators can then wonder whether norepinephrine still exerts a positive effect on myocardial contractility via the increase in DAP, despite an alteration of the β1-adrenergic pathway.

To answer this question, the investigators proposed to evaluate the effects of norepinephrine by TTE on cardiac contractility after the initial phase.

DETAILED DESCRIPTION:
Patients presenting with septic shock for 24 hours or more and meeting the inclusion criteria may be included.

The course of the study will be as follows:

T0: collection (as part of usual care) of clinical circulatory parameters (heart rate, systolic/diastolic/mean blood pressure) and biological parameters (arterial lactate and ScVo2) and performance of echocardiography.

Parameters collected during TTE:

* Concerning the main judgment criterion and the secondary judgment criteria:

  * Left ventricular ejection fraction (LVEF) by the Simpson Biplane method,
  * Cardiac output and cardiac index by continuity equation (measurement of left ventricular outflow chamber (mm) and sub-aortic time-velocity integral (cm/s)).
  * Tricuspid Annular Systolic Excursion (TAPSE) (mm)
  * S wave at the tricuspid ring (cm/s)
* Other parameters collected systematically:

  * Surface of the left ventricle (end-systolic and end-diastolic),
  * Global strain of the left ventricle
  * Mitral Annular Plane Systolic Excursion (MAPSE) (mm)
  * Left ventricular filling pressure (LVRP) (at the mitral annulus, E, A, e', S' waves, E/A ratio, E/e');
  * Maximum tricuspid regurgitation velocity (m/s) to estimate systolic pulmonary arterial pressure (PAPs) (mmHg)

T1: After the clinician in charge introduces or increases norepinephrine to achieve MAP ≥ 65mmHg, T1 will be when the goal of MAP ≥ 65mmHg is reached. This will be the target MAP for the management of septic shock of the patient in question according to the recommendations of learned societies.

Collection of clinical and biological circulatory parameters and performance of the TTE. The parameters collected will be the same as at T0.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years old
* Septic shock after 24 hours from its diagnosis
* MAP<65 mmHg for which the physician in charge decided to increase NE

Exclusion Criteria:

* Patient under Dobutamine
* Pregnancy
* Do not resuscitation decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from septic shock, after 24 hours of their diagnosis. Presenting with Mean arterial pressure (MAP)<65 mmHg or the target MAP For whom the physician in charge decided to increase the norepinephrine dose
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-03-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
The effect of the increase of Norepinephrine dose after restoring MAP on cardiac contractility evaluated by TTE : the left ventricular ejection fraction | through study completion, an average of 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided